CLINICAL TRIAL: NCT07031843
Title: Exploration of a Novel Prognostic Prediction Model for Liver Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: Juan Kang (Other)
Responsible Party: Sponsor-Investigator, Juan Kang, associate professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2025-078
Record Dates: First submitted 2025-06-19; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Cirrhosis
Keywords: cirrhosis; disease prognosis model; metabolomics; nutritional assessment
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with cirrhosis: A diagnosis of liver cirrhosis that meets the reference criteria of the Chinese Society of Hepatology's "Guidelines for the Diagnosis and Treatment of Liver Cirrhosis".

SUMMARY:
The liver, a key organ for metabolism and synthesis, is involved in protein, fat, and carbohydrate metabolism, as well as energy production. Hepatic injury and functional decline can lead to metabolic abnormalities in these three major nutrients, as well as in vitamins and trace elements. Malnutrition, one of the most common complications in cirrhosis patients, has a broader impact than traditional complications like hepatic encephalopathy, esophageal variceal bleeding, refractory ascites, and spontaneous bacterial peritonitis. It is closely related to patient prognosis. Therefore, malnutrition should be considered as important as ascites and hepatic encephalopathy in diagnosis and treatment, and nutritional metabolism should be incorporated into prognostic prediction models or scoring systems for cirrhosis patients.

Currently, the nutrition assessment of cirrhosis patients mostly uses relatively subjective methods such as scales and scores. There is no specific gold-standard diagnostic criterion for malnutrition in cirrhosis patients. Also, existing prognostic models for cirrhosis patients do not adequately consider the impact of nutritional factors on disease prognosis. Metabolomics technology can detect changes in the types and levels of nutritional metabolites in cirrhosis patients and analyze the differences in nutritional metabolites under various nutritional statuses and their relationship with the prognosis of cirrhosis patients. This helps objectively reveal the predictive value of nutrition metabolism for the prognosis of cirrhosis patients. However, metabolomics has been rarely used in nutrition assessment studies of cirrhosis patients and merits further research.

This study will employ a prospective cohort study design to analyze the baseline nutritional status of patients with liver cirrhosis, investigate the impact of nutritional factors on long-term prognosis, and develop a prognostic prediction model for liver cirrhosis that incorporates nutritional parameters.

DETAILED DESCRIPTION:
Patients with cirrhosis attending the Second Affiliated Hospital of Chongqing Medical University were included in this prospective study. Eligible subjects were determined based on the inclusion and exclusion criteria. Clinical data were collected, including gender, age, blood routine, liver and kidney function, coagulation function, comorbidities, complications, and disease progression. Various indicators were calculated, including body mass index (BMI), Prognostic Nutritional Index (PNI), Geriatric Nutritional Risk Index (GNRI), Model for End-Stage Liver Disease (MELD) score, MELD-Na score, and MELD 3.0 score. Nutritional risk screening and malnutrition assessment were also performed. Resting energy expenditure was measured by professionals, and blood samples were collected for non-targeted nutritional metabolite profiling. Patients were followed up at 3 months, 6 months, 1 year, and 2 years to assess survival status, hepatic adverse events, and complication occurrence. Statistical analysis was conducted to identify nutritional scores, indicators, or differential metabolite levels closely associated with patient prognosis. Variables for model construction and scoring were determined, assigned scores, and a novel prognostic prediction model for cirrhosis patients was developed and optimized. This study aims to integrate nutritional assessment into the prognostic evaluation system for cirrhosis patients, establishing a more objective, accurate, and comprehensive model. It provides evidence for nutritional intervention and improving patient prognosis and lays a foundation for further research. Additionally, metabolomics analysis of differential metabolites in cirrhosis patients with varying nutritional statuses and prognoses offers insights into the molecular mechanisms of nutritional metabolism's impact on prognosis.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for this study.

1. Willingness and ability to sign the informed consent form.
2. Male or female, aged 18 to 75 years.
3. A diagnosis of liver cirrhosis that meets the reference criteria of the Chinese Society of Hepatology's "Guidelines for the Diagnosis and Treatment of Liver Cirrhosis".
4. An expected survival of over 3 months.
5. Full civil competence.

Exclusion Criteria:

1. Primary liver cancer diagnosis, or supporting evidence of elevated alpha-fetoprotein (AFP≥100μg/L) for >3 months, or imaging evidence of hepatic cancer nodules.
2. Malignancy history within 5 years before screening, except for specific cured cancers (e.g., basal cell skin cancer); current or past major illnesses (as defined by the China Insurance Regulatory Commission's 25 critical illnesses) that may affect treatment, assessment, or compliance.
3. Severe pulmonary, cardiac, diabetic, or genetic metabolic diseases.
4. Psychiatric hospitalization, suicide attempts, or temporary disability due to mental illness in the past 5 years.
5. Pregnant or breastfeeding women.
6. Individuals deemed unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with liver cirrhosis in accordance with the reference criteria of the Chinese Society of Hepatology's "Guidelines for the Diagnosis and Treatment of Liver Cirrhosis".
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Death | From February 2023 to December 2026
  Death due to cirrhosis progression

SECONDARY OUTCOMES:
complication | From February 2023 to December 2026
  complication such as infection，ascites

CONTACTS AND LOCATIONS:
Overall Officials: juan Kang, M.D., Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China